CLINICAL TRIAL: NCT02183025
Title: Double Blind Study to Evaluate Efficacy and Safety of Meloxicam 7.5 mg and 15 mg Versus Mefenamic Acid 1500 mg in the Treatment of Dysmenorrhea
Brief Title: Efficacy and Safety Study of Meloxicam Versus Mefenamic Acid in Patients With Dysmenorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107.191
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Meloxicam; Mefenamic Acid

ARMS (3):
- Meloxicam 7.5 mg (Experimental)
  Interventions: Drug: Meloxicam 7.5 mg; Drug: Placebo matching 15 mg meloxicam; Drug: Placebo matching 500 mg mefenamic acid
- Meloxicam 15 mg (Experimental)
  Interventions: Drug: Meloxicam 15 mg; Drug: Placebo matching 7.5 mg meloxicam; Drug: Placebo matching 500 mg mefenamic acid
- Mefenamic acid 1500 mg (Active Comparator): 500 mg three times daily
  Interventions: Drug: Mefenamic acid 500 mg; Drug: Placebo matching 7.5 mg meloxicam; Drug: Placebo matching 15 mg meloxicam

INTERVENTIONS:
Drug: Meloxicam 7.5 mg
  Arms: Meloxicam 7.5 mg
Drug: Meloxicam 15 mg
  Arms: Meloxicam 15 mg
Drug: Mefenamic acid 500 mg
  Arms: Mefenamic acid 1500 mg
Drug: Placebo matching 7.5 mg meloxicam
  Arms: Mefenamic acid 1500 mg; Meloxicam 15 mg
Drug: Placebo matching 15 mg meloxicam
  Arms: Mefenamic acid 1500 mg; Meloxicam 7.5 mg
Drug: Placebo matching 500 mg mefenamic acid
  Arms: Meloxicam 15 mg; Meloxicam 7.5 mg

SUMMARY:
To access the efficacy and safety of Meloxicam 7.5 mg and 15 mg once daily compared with Mefenamic acid 500 mg t.i.d. over a treatment period of 3-5 days, during an observation period of 3 menstrual cycles, for the symptomatic relief of primary dysmenorrhea

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 to 40 years
* Patients experiencing primary (functional) dysmenorrhea during the last 3 consecutive menstrual periods. Diagnosis will be based on symptoms and clinical signs: abdominopelvic pain, may radiate to the back and along the thighs; systemic symptoms including nausea, vomit, diarrhoea, headache, fatigue, nervousness, dizziness; the symptomatology should be usually some hours to one day before commencement of visible vaginal bleeding
* Evaluation of lumbar and/or abdominopelvic pain due to dysmenorrhea > 35 mm through a 100 mm visual analogue scale (VAS)
* Outpatients
* Patients granting their written informed consent
* Therapy with a NSAID (nonsteroidal antiinflammatory drug) is required or recommended

Exclusion Criteria:

* Known or suspected hypersensitivity to trial drugs or their excipients, analgesics, antipyretics or NASIDs
* Analgesic concomitant treatment (between each cycle paracetamol administration will be allowed)
* To initiate hormonal contraception or intrauterine devices after inclusion to this trial or during the last 3 months
* Abdominal surgery or pelvic procedure scheduled during the study
* Patients with organic dysmenorrhea (endometriosis, salpingitis, adnexitis, uterine retroversion, tubal cysts, ovarian cysts, pathological vaginal secretion, painful pelvic exploration, etc.)
* Patients with neoplastic disorders
* History of recent abdominal or pelvic trauma requiring surgery
* Peptic ulcer within the past 6 months
* Pregnancy or breast feeding
* Asthma, nasal polyps, angioneurotic edema or rash following aspirin or NSAIDs administration
* Concomitant treatment with anti-coagulants, including heparin and aspirin, lithium or methotrexate
* Concomitant administration of other NSAIDs (including aspirin > 150 mg daily) or analgesics
* Confinement to bed rest
* Administration of any NSAID during two days (three for oxicams) before the first administration of the trial drug
* Present treatment or treatment within the last two months with corticosteroids
* Impaired renal function (serum urea > 125 % of the upper limit of normal range; serum creatinine > 150 % of the upper limit of normal range)
* Sever liver injury (alanine amino transferase ALAT > 2 x the upper normal range limit or aspartate amino transferase ASAT > 2 x the upper normal range limit)
* Hematological disorder (platelet count < 100,000/mm**3, leucocyte count < 3,000/mm**3)
* Participation in another clinical trial during this study or the previous month
* Previous participation in this trial
* Patient unable to comply with protocol
* Bleeding disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 337 (Actual)
Dates: Start 1998-01; Primary Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of severity of lumbar and/or abdominal pain on a visual analogue scale (VAS) | Baseline and day 3-5 of each treatment cycle

SECONDARY OUTCOMES:
Final global assessment of efficacy by patient on a 4-point scale | day 3-5 of the second treatment cycle
Final global assessment of efficacy by investigator on a 4-point scale | day 3-5 of the second treatment cycle
Final global assessment of tolerability by patient on a 4-point scale | day 3-5 of the second treatment cycle
Final global assessment of tolerability by investigator on a 4-point scale | day 3-5 of the second treatment cycle
Number of Participants with Adverse Events (AE) | Up to 4 weeks after last treatment cycle
Incidence of significant laboratory events | Up to 4 weeks after last treatment cycle
Number of perforations, ulcerations and/or bleedings (PUB) of the upper gastro-intestinal tract | Up to 4 weeks after last treatment cycle
Number of gastro-intestinal adverse events (GI-AEs) | Up to 4 weeks after last treatment cycle
Duration of hospitalization stay due to GI-AEs | Up to 4 weeks after last treatment cycle
Number of additional visits at physician due to GI-AEs | Up to 4 weeks after last treatment cycle
Duration of hospitalization due to drug related AEs | Up to 4 weeks after last treatment cycle
Number of withdrawals due to AEs | Up to 4 weeks after last treatment cycle
Intensity of AEs on a 3-point scale | Up to 4 weeks after last treatment cycle
Evaluation of labor and/or daily life disability associated with dysmenorrhea on a VAS | Baseline and day 3-5 of each treatment cycle
Change in severity of symptomatology associated with dysmenorrhea | Baseline and day 3-5 of each treatment cycle